CLINICAL TRIAL: NCT01920607
Title: Medical and Economic Evaluation of a Magnetic Anal Sphincter for Patients With Severe Anal Incontinence
Acronym: MOS STIC
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC13_0209
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Fecal Incontinence; Anal Incontinence
Keywords: Fecal Incontinence.; Anal Incontinence.; Functional Bowel Disorders.; SNS.; Artificial Sphincters.; Magnetic Anal Sphincter.
MeSH Terms: conditions — Fecal Incontinence; Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NMS (Active Comparator): Implantation under general of local anesthesia of sacral nerve stimulation system (Interstim Therapy)
  Interventions: Device: sacral nerve stimulation
- SAM (Experimental): Implantation under general anesthesia of magnetic anal sphincter (Fenix)
  Interventions: Device: magnetic anal sphincter

INTERVENTIONS:
Device: magnetic anal sphincter
  Other Names: Fenix
  Arms: SAM
Device: sacral nerve stimulation
  Other Names: Interstim
  Arms: NMS

SUMMARY:
The purpose of this study is to compare 2 surgical treatments of severe fecal incontinence (defined as more than a major leak per week). The hypothesis of this "non-inferiority" trial is that magnetic anal sphincter is clinically as effective as SNS, but more cost-effective in managing fecal incontinence

DETAILED DESCRIPTION:
Severe anal incontinence, defined as the uncontrolled passing of stool at least once a week, is a problem that has a serious impact on the quality of life. In the event of failure of conservative treatments, surgery can help improve continence problems in a significant number of cases.

Sacral nerve stimulation is currently the standard surgical treatment for severe anal incontinence when sphincter repair (sphincteroplasty) is not recommended.

A new method of treatment based on sphincter reinforcement through the implanting of a band of magnetic beads*, has proved to be reliable and efficient on a small series of cases, particularly after the failure of sacral nerve stimulation.

The aim of our trial, which compares the "magnetic anal sphincter* and sacral nerve stimulation" in a homogeneous population of patients affected by severe anal incontinence is to define the position of this new approach in the treatment algorithm of this functional disorder, determining its clinical and medical/economic advantages compared to those of the current standard treatment.

* FenixTM (Torax Medical)

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (male or female) of 18 to 75 years of age
* Affected by severe anal incontinence (SAI)*.
* Documented failure of conservative treatment (reeducation and medical treatment)
* With functional anal sphincter**
* Agrees to take part in the study and has signed the informed consent form
* Agrees to undergo post-operative surveillance for a period of one (1) year
* Covered by National Insurance

  * Defined as follows: at least one involuntary passing of stool per week measured by collecting data on incontinence accidents on a 3-week stool record chart, with the continence problem developing over more than 6 months. **Defined as follows: external sphincter intact (without injury or after sphincter repair) or external sphincter altered, with an injury of a size that does not justify sphincter repair.

Internal sphincter injuries not taken into account (by professional consensus).

Exclusion Criteria:

* Anorectal or pelvic malformations
* Local conditions incompatible with the proposed sizes of the MAS (extreme obesity, thickness of the tissue in the anorectal area)
* Sequelae of rectal resections - presence of cancer of the rectum or anus
* Rectal prolapse and/or major pelvic floor disorders
* Major chronic disorder of the intestinal motility, irritable bowel syndrome, repeated faecalomas, megarectum
* Extensive sphincter degeneration
* Consequences of radiation-induced rectitis and chronic inflammatory diseases of the bowel (Crohn's disease)
* Neurological disorders or systemic diseases (multiple sclerosis, scleroderma, paraplegia)
* Festering sores of the perineal and/or anorectal regions
* Known or suspected risks of allergy to titanium
* Active pelvic infection
* Contraindications to SNS:

  * Cardiac stimulator or defibrillator implant
  * Malformation of the sacrum
  * Patient exposed to Magnetic Resonance Imaging
  * Skin diseases exposing the patient to the risk of infection (at the investigator's discretion)
  * Patient scheduled for diathermy or ablation by radiofrequency
* Pregnant women
* Adults under guardianship
* Patients involved in a mobility project in the year following the operation
* Patient already subjected to one or other of the therapeutic approaches (MAS or SNS) Please note: coagulation problems (including anti-aggregant or anti-coagulant treatments) are not a contraindication if these problems can be corrected during the perioperative period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Average number of fecal incontinence episodes | 6 months
  Average number of fecal incontinence episodes per week over a period of 3 weeks, 6 months after the implantation of a magnetic anal sphincter (FenixTM magnetic anal sphincter group) or of the Spinelli electrode during the PNE test (sacral nerve stimulation group), on the basis of a standardised stool diary

SECONDARY OUTCOMES:
Overall cost for the health care system | 12 months
  Overall cost for the health care system including implantation and follow-up - Duration and cost of hospital admissions,- Cost of covering any complications arising
Respective complications of the two therapeutic approaches | 12 months
  Number and nature of the complications over 12 months, according to the Clavien-Dindo classification
Functional results at 6 and 12 months, compared with baseline | Baseline, 6 & 12 months
  Stool record chart, faecal incontinence score (Wexner), recourse to antidiarrhoeal treatment, the taking of analgesics, constipation score (ODS), recourse to a treatment for constipation
Quality of life and overall satisfaction | Baselnie, 6 & 12 months
  Quality of life and overall satisfaction of the patient at 6 and 12 months, compared with baseline:Quality of life score specific to faecal incontinence (FIQL), General quality of life scores (SF 36 and EQ-5D)
Anorectal manometry data | Baseline & 6 months
  Sphincter pressure at rest, voluntary contractions, rectal maximum tolerable volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Background] Wong MT, Meurette G, Wyart V, Lehur PA. Does the magnetic anal sphincter device compare favourably with sacral nerve stimulation in the management of faecal incontinence? Colorectal Dis. 2012 Jun;14(6):e323-9. doi: 10.1111/j.1463-1318.2012.02995.x. PMID 22339789